CLINICAL TRIAL: NCT06459193
Title: Evaluation of Trimetazidine in Alleviating Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: Trimetazidine Efficacy in Attenuating Paclitaxel-Induced Peripheral Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Asmaa Najm Iqbal Ahmed, Demonstrator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2301006
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
Keywords: Paclitaxel; Trimetazidine; quality of life; nerve growth factor; peripheral neuropathy
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Peripheral Nervous System Diseases | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Trimetazidine Tablet 35 mg once daily for the treatment period
  Interventions: Drug: Trimetazidine
- Control (Placebo Comparator): Placebo once daily for the treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimetazidine — Trimetazidine 35 mg tab once daily
  Arms: Intervention
Drug: Placebo — Placebo once daily
  Arms: Control

SUMMARY:
This proof-of-concept study evaluated the effect of Trimetazidine on the incidence of paclitaxel-induced peripheral neuropathy in patients with breast cancer.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a major adverse effect of many commonly used chemotherapeutic agents that greatly affect patient quality of life. Paclitaxel (PTX), one of the main neurotoxic classes of anticancer drugs, is used to treat several types of solid tumors, including breast cancer. Development of PTX-induced peripheral neuropathy (PIPN) during cancer treatment requires dose reduction limiting its clinical benefits.

The only currently recognized prophylactic measure for chemotherapy-induced peripheral neuropathy (CIPN) is monitoring for pre-existing neuropathies and then the early detection of clinical symptoms of neuropathy in subjects undergoing neurotoxic chemotherapy treatment.

Preclinical data has shown that the neuroprotective effect of trimetazidine (TMZ) can attenuate PIPN.

TMZ has preclinical evidence about its preventive capacity against peripheral neuropathy. Which represents a possible prophylactic strategy for attenuating PIPN. TMZ is commercially available in various preparations that are relatively affordable and well-tolerated, making it a valid candidate for clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who will receive paclitaxel.
* Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
* Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count≥100,000/mm3), liver function (serum total bilirubin <1.5 mg/dl), renal function (creatinine < 1.5 mg/dl).

Exclusion Criteria:

* Patients with signs and symptoms of clinical neuropathy at baseline.
* Patients with diabetes mellitus, alcoholic disease, heart failure, pregnant or lactating women.
* Patients receiving vitamin/ supplementation drugs that interfere with the study intervention.
* Patients with contraindications to trimetazidine including Parkinson's disease, Parkinsonian symptoms, tremors, restless leg syndrome, and other related movement disorders.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-23 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of chemotherapy induced-peripheral neuropathy using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria | weekly for up to 8 weeks
  Number of patients reported neuropathy from paclitaxel. a 1 to 5 graded scale; where grade (1) is the minimum value and grade (5) is the maximum value, a greater grades mean greater symptomatic burden.
Patient's Quality of Life | at baseline, at the end of 4 weeks and at the end of 8 weeks
  measures the quality of life using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity FACT/GOG-NTX (Version 4) questionnaire.
  A total score ranging from 0 (minimum value) to 44 (maximum value), where lower scores mean greater symptomatic burden.

SECONDARY OUTCOMES:
Changes in serum levels of biomarker namely nerve growth factor (NGF). | at baseline and at end of 8 weeks
  measuring serum level of nerve growth factor using enzyme-linked immunoassay (ELISA) Kit.
Adverse effects of using trimetazidine in preventing Paclitaxel Induced Peripheral Neuropathy. | at baseline and weekly up to 8 week
  any adverse/ side effect will be evaluated.
Severity of chemotherapy induced-peripheral neuropathy. | at baseline, at the end of 4 weeks and at the end of 8 weeks
  The severity of paclitaxel-induced peripheral neuropathy using VAS visual analogue scale.
  a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa N. Iqbal Ahmed, Demonstrator, Principal Investigator — Clinical Pharmacy Department, Faculty of Pharmacy, Minia University, Minia, Egypt.; Engy A. Wahsh, Asst. Prof., Study Director — Clinical Pharmacy Department, Faculty of Pharmacy, October 6 University, Giza, Egypt; Fatma M. Mady, Professor, Study Chair — Pharmaceutics department, Faculty of Pharmacy, Minia University, Minia, Egypt.; Eman M. Sadek, Lecturer, Study Director — Clinical pharmacy Department, Faculty of Pharmacy, Minia University, Minia, Egypt.; Ahmed Mostafa Abd-Elaziz, Lecturer, Study Director — Department of Clinical Oncology, Faculty of Medicine, Minia University, Minia, Egypt.; Noha Mahmood Abd-Allah, Lecturer, Study Director — Department of Clinical Pathology, Faculty of Medicine, Minia University, Minia, Egypt.
Locations (1):
- Minia Oncology Center, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalefa HG, Shawki MA, Aboelhassan R, El Wakeel LM. Evaluation of the effect of N-acetylcysteine on the prevention and amelioration of paclitaxel-induced peripheral neuropathy in breast cancer patients: a randomized controlled study. Breast Cancer Res Treat. 2020 Aug;183(1):117-125. doi: 10.1007/s10549-020-05762-8. Epub 2020 Jun 29. PMID 32601973
- [Background] Haroun EA, Mansour NO, Eltantawy A, Shams MEE. Effect of cilostazol on preventing paclitaxel-induced neuropathy in patients with breast cancer: A randomized controlled trial. Pharmacotherapy. 2023 Sep;43(9):872-882. doi: 10.1002/phar.2830. Epub 2023 Jun 12. PMID 37199288
- [Background] Hammad ASA, Sayed-Ahmed MM, Abdel Hafez SMN, Ibrahim ARN, Khalifa MMA, El-Daly M. Trimetazidine alleviates paclitaxel-induced peripheral neuropathy through modulation of TLR4/p38/NF-kappaB and klotho protein expression. Chem Biol Interact. 2023 May 1;376:110446. doi: 10.1016/j.cbi.2023.110446. Epub 2023 Mar 9. PMID 36898573